CLINICAL TRIAL: NCT00028210
Title: Enhancement of Tactile Spatial Acuity in Upper Limb Amputees
Brief Title: Enhanced Tactile (Touch) Spatial Acuity in Upper Limb Amputees
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020067; 02-N-0067
Record Dates: First submitted 2001-12-17; First posted 2001-12-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Amputation
Keywords: Amputee; Plasticity; Somatosensory; Upper Limb Amputation; Tactile Performance; Cortical Reorganization; Healthy Volunteer; HV; Normal Control

SUMMARY:
This study will examine whether tactile (touch) abilities at the lip are more acute in people with upper limb amputation compared with healthy normal volunteers. People with an amputated upper limb have an expanded brain representation of the lip that may correlate with heightened tactile spatial acuity.

Normal volunteers will be recruited for this study. Candidates will be screened with physical and neurological examinations. (Amputee volunteers will be studied at the amputee clinic at the University of Tubingen, Germany.)

Participants will sit comfortably in a chair, wearing a blindfold, during the following experiments:

* Plastic domes with grooves are placed on parts of the lower lip on either side for a few seconds. The volunteer is then asked to identify the direction of the grooves relative to the long axis of the lip.
* The participant's arm is placed in a cast and the index finger is immobilized. The same test done on the lip is repeated on the distal part of the index finger.

Each part of the test lasts about 20 minutes, and the entire experiment takes about 2 hours.

DETAILED DESCRIPTION:
Upper limb amputation leads to expansion of the cortical representation of the lip into the adjacent deafferented hand representation. It is conceivable that this enlargement of the lip representation may translate into a behavioral gain. The purpose of this protocol is to test the hypothesis that upper limb amputation in humans results in higher tactile spatial acuity at the lip. This would represent the first demonstration of chronic deafferentation-induced behavioral gains within the somatosensory system.

ELIGIBILITY:
INCLUSION CRITERIA:

Normal volunteers who are willing and able to stay relaxed and collaborative for a period of up to 2 hours.

Subjects with upper limb amputation more than one year before testing.

EXCLUSION CRITERIA:

Neurological or psychiatric disease

Excessive callus at the palm of the fingers

Subjects, who are unable to perform or understand the task

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2001-12; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Elbert T, Flor H, Birbaumer N, Knecht S, Hampson S, Larbig W, Taub E. Extensive reorganization of the somatosensory cortex in adult humans after nervous system injury. Neuroreport. 1994 Dec 20;5(18):2593-7. doi: 10.1097/00001756-199412000-00047. PMID 7696611
- [Background] Flor H, Elbert T, Knecht S, Wienbruch C, Pantev C, Birbaumer N, Larbig W, Taub E. Phantom-limb pain as a perceptual correlate of cortical reorganization following arm amputation. Nature. 1995 Jun 8;375(6531):482-4. doi: 10.1038/375482a0. PMID 7777055
- [Background] Kaas JH, Merzenich MM, Killackey HP. The reorganization of somatosensory cortex following peripheral nerve damage in adult and developing mammals. Annu Rev Neurosci. 1983;6:325-56. doi: 10.1146/annurev.ne.06.030183.001545. No abstract available. PMID 6340591